CLINICAL TRIAL: NCT00097929
Title: A Phase II Clinical Trial of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Relapsed Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: An Investigational Drug Study With Suberoylanilide Hydroxamic Acid in Relapsed Diffuse Large B-cell Lymphoma (0683-013)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-013; MK0683-013; 2004_029; NCT00124631 (obsolete NCT alias)
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: B-cell Lymphoma
Keywords: Relapsed Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Vorinostat; Duration of Therapy

INTERVENTIONS:
Drug: MK0683, vorinostat, Suberoylanilide Hydroxamic Acid (SAHA) / Duration of Treatment 6 Months

SUMMARY:
A study to determine the safety, tolerability, and anti-tumor effectiveness of an oral investigational drug in the treatment of relapsed diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older with relapsed Diffuse Large B-cell Lymphoma (DLBCL).
* Stable disease or better for at least 3 months on most recent treatment
* Have not received any chemotherapy, radiation therapy, major surgery, or any other investigational therapy for at least 4 weeks prior to entry in this study
* Adequate blood testing, liver, and kidney function as required by the study.
* Eligible subjects will allow tissue samples to be examined and stored.

Exclusion Criteria:

* Patient has been treated with other investigational agents with a similar anti-tumor mechanism.
* Patient should not have failed more than 3 prior treatment regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2006-07-31 (Actual); Study Completion 2006-07-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate based on FDG-PET and CT scan findings.

SECONDARY OUTCOMES:
Response duration, Progression-free survival, Time to progression, Time to response, 3-Month and 6-month progression free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Crump M, Coiffier B, Jacobsen ED, Sun L, Ricker JL, Xie H, Frankel SR, Randolph SS, Cheson BD. Phase II trial of oral vorinostat (suberoylanilide hydroxamic acid) in relapsed diffuse large-B-cell lymphoma. Ann Oncol. 2008 May;19(5):964-9. doi: 10.1093/annonc/mdn031. Epub 2008 Feb 21. PMID 18296419
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html